CLINICAL TRIAL: NCT06775041
Title: A Phase 2a, Randomized, Open-Label Study to Determine the Optimal Dose and Evaluate the Safety, Tolerability, and Pharmacokinetics of Progerinin in Patients With Hutchinson-Gilford Progeria Syndrome (HGPS)
Brief Title: Study to Determine Optimal Dose and Evaluate Safety, Tolerability, and Pharmacokinetics of Progerinin in Patients With Hutchinson-Gilford Progeria Syndrome (HGPS)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: PRG Science & Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRG-PRO-005
Record Dates: First submitted 2024-12-11; First posted 2025-01-14 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Hutchinson-Gilford Progeria Syndrome
MeSH Terms: conditions — Progeria | interventions — lonafarnib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Progerinin + Lonafarnib (Experimental): Subjects who have successfully completed the Screening phase will enter the treatment phase of the study and be randomized to a treatment arm. Subjects randomized to the progerinin + lonafarnib arm will take progerinin at a dose dependent on their body weight and will continue taking lonafarnib per the package insert.
  For each dose cohort, subjects will complete a 28-day treatment period of toxicity assessment, and a minimum four-month treatment period for plasma progerin evaluation. After the last subject completes the toxicity assessment period, the independent Data Monitoring Committee (iDMC) will meet to confirm that subjects can be escalated to the next dose. All subjects will remain on the current dose until the iDMC decision is confirmed. Each subject will only be escalated to the next dose after their 4-month (±2 weeks) plasma progerin sample is collected.
  Interventions: Drug: Progerinin; Drug: Lonafarnib
- Lonafarnib Naïve (Other): Subjects with no prior treatment with lonafarnib (i.e., no commercial or managed access program source) may be enrolled to initiate treatment with lonafarnib monotherapy. These subjects will initiate lonafarnib therapy in preparation for an upcoming phase of the study following the completion of phase 2a. These subjects will be excluded from the analysis of this phase 2a study. They will come to the study site for a baseline visit and at one year for assessment as described later in this protocol.
  Interventions: Drug: Lonafarnib
- Lonafarnib (Active Comparator): Subjects in the main study arms (Progerinin + Lonafarnib and non-naïve Lonafarnib) will continue taking lonafarnib per the package insert. Subjects randomized to the lonafarnib alone arm will not take progerinin during this study.
  Interventions: Drug: Lonafarnib

INTERVENTIONS:
Drug: Progerinin — Dosing will be determined based on body weight. Dosing ranges from 500mg to 1500mg daily. Progerinin is available in sachets of 250 mg or 350 mg for oral use.
  Arms: Progerinin + Lonafarnib
Drug: Lonafarnib — Lonafarnib is considered as the standard of care (SOC). Subjects in the randomized arms will continue taking lonafarnib per the package insert. Subjects in the lonafarnib naïve arm will initiate lonafarnib as per FDA-approved study 07-01-7505.

SUMMARY:
Researchers will compare treatment with progerinin plus lonafarnib vs lonafarnib alone to assess optimal dosing, safety, tolerability, and pharmacokinetics in patients with Hutchinson-Gilford Progeria Syndrome (HGPS). Subjects in the randomized study arms will continue to take the standard of care (SOC), lonafarnib, and will be randomized to either take SOC alone or in combination with progerinin.

DETAILED DESCRIPTION:
During this trial, a total of 10 subjects will be randomized in a 4:1 ratio to receive treatment with progerinin plus lonafarnib vs lonafarnib alone. Dose escalation will occur through intra-subject dose titration. Two ascending doses of progerinin will be assessed. The dose levels proposed in this study were determined using body weight based on adult doses assessed in previously completed studies, and on a simulated population pharmacokinetic (PK) model. If systemic exposures of Progerinin in pediatric patients are lower than those in adults, a dose escalation may be added at the end of the study.

Progerinin will be administered, with food. The study treatment is available in sachets of 250 mg or 350 mg and the doses in the study range from 500 to 1500 mg daily, dosed BID (twice a day).

Lonafarnib is considered as the standard of care (SOC) and all subjects in the randomized study arms will continue taking lonafarnib for the duration of the study. Subjects who are not already taking lonafarnib will also have the opportunity to initiate lonafarnib on this study as part of the lonafarnib naïve arm (separate from the randomized study arms).

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible for enrollment in the study only if they meet ALL the following criteria at time of Screening:

1. Subjects ≥ 1 year of age and weight ≥ 17.6 lb (8 kg).
2. Subject must have confirmatory mutational analysis showing the classic HGPS mutation (c. 1824 C>T), nonclassic HGPS, Zmpset24 gene mutation, or other LMNA mutation (all subjects will havedocumentation of genetic testing prior to enrollment). *Only subjects with progerin producing mutations will be eligible for randomization. Other PL are eligible to enroll as naïve subjects (see note for criterion #5).
3. Subject must display clinical signs of Progeria as per the clinical trial team.
4. Subject must be willing and able to come to Boston for appropriate assessments and examinations.
5. Subject must be taking lonafarnib for at least 4 months prior to enrollment and have no history of grade 3 or 4 side effects that can be probably or possibly attributed to lonafarnib for at least 2 months prior to enrollment.

   Note: Subjects with no prior treatment (i.e., no commercial or managed access program source) with lonafarnib may be enrolled to initiate treatment with lonafarnib monotherapy. These subjects will initiate lonafarnib therapy in preparation for an upcoming phase of the study following the completion of phase 2a. These subjects will be excluded from the analysis of this phase 2a study. These subjects must be at least 12 months of age per lonafarnib package insert.
6. Subjects must have had no recent fractures or major surgery (within four weeks).
7. Subject must have adequate organ and marrow function as defined by the following parameters:

   1. Blood: APC (ANC + bands + monocytes) >1,000/µL, platelets >75,000/µL (transfusion independent); hemoglobin >9 g/dL.
   2. Renal: creatinine ≤ 1.5 times normal for age or Glomerular Filtration Rate (GFR) >70 mL/min/1.73m2.
   3. Hepatic: bilirubin ≤1.5x upper limit of normal for age; Serum Glutamic Pyruvic Transaminase (SGPT) (Alanine Transaminase, [ALT]) < and Serum Glutamic-Oxaloacetic Transaminase (SGOT) (Aspartate Aminotransferase, [AST]) ≤ 2.5x normal range for age.
8. The subject is willing to provide written informed assent form, when possible, to participate in the study after reading the informed assent form and the information provided and has had the opportunity to discuss the study with the investigator or designee. Additionally, the subject's legally authorized guardian (LAR) is willing to provide written informed consent.
9. The subject is able to communicate satisfactorily with the investigator and to participate in, and comply with, the requirements of the study.
10. The subject (or LAR) is able to understand the nature of the study and any potential hazards associated with participating in it.
11. Negative pregnancy test for female subjects of childbearing potential and those who have not been surgically sterilized or who do not have verbal or laboratory confirmation of two years postmenopausal status. Women of childbearing potential (WOCBP) and Women of non-childbearing potential are eligible to participate. Women of childbearing potential should use an acceptable method of birth control and agree to continue to use this method for the duration of the study and for 90 days after taking the last dose of Progerinin.

Acceptable methods of contraception include abstinence, female subject/partner's use of hormonal contraceptive (oral, implanted, or injected) in conjunction with a barrier method (WOCBP only) (e.g., diaphragm, cervical cap, male condom, and female condom and spermicidal foam, sponges, and film), female subject/partner's use of an intrauterine device (IUD), or if the female subject/partner is surgically sterile (e.g., bilateral tubal ligation, hysterectomy) or two years postmenopausal at time of screening. All male subjects/partners (excluding men who have been sterilized) must agree to consistently and correctly use a condom for the duration of the study and for 90 days after taking the study drug. In addition, subjects may not donate sperm for the duration of the study and for 90 days after taking study drug.

Exclusion Criteria:

Subjects meeting ANY of the following criteria at time of Screening will be excluded from enrollment:

1. Other than the drugs used in this protocol, other drugs targeted to treat Progeria are excluded. Drugs to treat symptoms of Progeria are permitted.
2. Subjects are taking medications that significantly affect the metabolism of Progerinin.
3. Subjects with an active bleeding diathesis or on oral anti-vitamin K medication (except low dose coumadin).
4. Subjects who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

   1. known severely impaired lung function
   2. active (acute or chronic) or uncontrolled severe infections.
   3. liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis.
   4. history of hepatitis B or hepatitis C documented by history and confirmed by serology if positive for history.
5. Other concurrent severe and/or uncontrolled medical disease that could compromise participation in the study (i.e., uncontrolled diabetes, uncontrolled hypertension, severe infection, severe malnutrition, chronic liver or renal disease, active upper GI tract ulceration).
6. A known history of Human Immunodeficiency Virus (HIV) seropositivity or known immunodeficiency.
7. Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of Progerinin (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection). A nasogastric tube (NG tube) or gastric tube (G tube) is allowed.
8. Subjects who have known or suspected hypersensitivity to any of the excipients included in the formulation should not be treated.
9. Subjects who have used marijuana or other (Tetrahydrocannabinol) THC containing products either recreationally or for medical purposes within three months prior to entering the study.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-01-13 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in plasma progerin concentration | Baseline and Month 4 of each cohort
Incidence of Dose Limiting Toxicities (DLTs) | From baseline to follow-up (approximately 13 months)
Incidence and severity of Treatment-Emergent Adverse Events (TEAEs) | From baseline to follow-up (approximately 13 months)
Incidence of withdrawals due to Adverse Events (AEs) | From baseline to follow-up (approximately 13 months)
Incidence of Treatment-Related Adverse Events | From baseline to follow-up (approximately 13 months)
Incidence of Serious Adverse Events (SAEs) | From baseline to follow-up (approximately 13 months)
Change/shifts in laboratory values from baseline | From baseline to follow-up (approximately 13 months)
Change in blood pressure from baseline | From baseline to follow-up (approximately 13 months)
Change in heart rate from baseline | From baseline to follow-up (approximately 13 months)
Change in respiratory rate from baseline | From baseline to follow-up (approximately 13 months)
Change in temperature from baseline | From baseline to follow-up (approximately 13 months)
Change in Electrocardiogram (ECG) parameter, ventricular rate (beats per minute), from baseline | From baseline to follow-up (approximately 13 months)
Change in Electrocardiogram (ECG) parameter, PR interval (msec), from baseline | From baseline to follow-up (approximately 13 months)
Change in Electrocardiogram (ECG) parameter, QRS interval (msec), from baseline | From baseline to follow-up (approximately 13 months)
Change in Electrocardiogram (ECG) parameter, QT interval (msec), from baseline | From baseline to follow-up (approximately 13 months)
Change in Electrocardiogram (ECG) parameter, QTc interval (msec), from baseline | From baseline to follow-up (approximately 13 months)
Maximum observed plasma drug concentration (Cmax) | Baseline, and pre-dose (0 hr) and 2-5 hr post-dose at Month 4 of each cohort
Apparent terminal elimination half-life (t1/2) | Baseline, and pre-dose (0 hr) and 2-5 hr post-dose at Month 4 of cohort1 & cohort 2
Time to maximum observed plasma drug concentration (Tmax) | Baseline, and pre-dose (0 hr) and 2-5 hr post-dose at Month 4 of cohort1 & cohort 2
Area under the plasma drug concentration-time curve (AUC) from time 0 to the end of the dosing period (AUC0-τ) | Baseline, and pre-dose (0 hr) and 2-5 hr post-dose at Month 4 of cohort1 & cohort 2
Clearance (CL) | Baseline, and pre-dose (0 hr) and 2-5 hr post-dose at Month 4 of cohort1 & cohort 2
Covariates: Age | Baseline, and pre-dose (0 hr) and 2-5 hr post-dose at Month 4 of each cohort
Covariates: Body weight | Baseline, and pre-dose (0 hr) and 2-5 hr post-dose at Month 4 of each cohort

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No